CLINICAL TRIAL: NCT00662402
Title: Impact of Extensive Consultation on Career Development Grant Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: K-Trial
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Career Development Grant Outcomes
Keywords: K Grant; Career Advancement; Award; Consultation; Application; K; The NIH priority score of the reviewed proposal.; Percent of subjects who obtain funding for proposal.; Percent of subjects who submit proposals for funding.
MeSH Terms: interventions — Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-Extensive Consultations (Experimental): Intervention- Receives extensive consulting services
  Interventions: Other: Extensive Consultations
- 2-Regular levels of service (No Intervention): Control - Receives regular levels of service; one hour free services from each of the 4 units, with option to pay for more.

INTERVENTIONS:
Other: Extensive Consultations — receives 15 free hours of multidisciplinary consultations towards the preparation of their career development grant.
  Other Names: Consultations; Extensive Multi-disciplinary Consultations
  Arms: 1-Extensive Consultations

SUMMARY:
In this study we wish is to determine whether extensive (up to 15 hours) multidisciplinary consultation in biostatistics, study design, data management, ethics, and writing provided by the UCSF Clinical and Translational Science Institute's (CTSI) Consultation Services program, improves peer review scores of career development grants compared to usual levels of consultation.

We hypothesize that extensive multidisciplinary consultation will improve peer review scores of career development grants compared to usual levels of consultation.

We hypothesize that extensive multidisciplinary consultation will lead to greater numbers of funded grants when compared to the usual levels of consultation.

DETAILED DESCRIPTION:
CTSI Consultation Services is one of the largest programs within the UCSF CTSI. It was created to improve the quality and efficiency of clinical and translational research through the provision of expert consultation. The program is divided into units that provide access to expert consultants in biostatistics, research design (with consultants representing multiple distinct methodologies and disease interests), data management (including data structure and database design), ethics, and scientific writing. With funding from the NIH, the program is able to offer a free hour of consultation in each of its units (up to 4 hours) but charges for additional services to cover costs.

There have been no studies of research consultation services. Though the benefit may seem self evident, such programs are expensive and distract senior researcher from more creative work. Justifying research consultation is important given the multitude of activities vying for attention and funding. Observational studies of the impact of research consultation services will always be limited by confounding, particularly confounding by indication since those seeking such services may be more highly motivated and organized. Thus, a randomized trial is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Applying for a Career Development grant from the NIH.
* Anticipated submission date is 3 or more months in the future
* Resident, fellow, or junior faculty member at UCSF or a CTSI-affiliated institution.
* Recognized potential benefit from additional consultation

  * Additional areas that could be improved as judged by the subject and the initial consultant
  * Adequate time to provide consultation before submission date

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2008-04; Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
NIH priority score of the reviewed proposal, with unsubmitted or unscored proposals counted as priority scores that are right-censored at 300 (old system) or 50 (new system) | 30 Months

SECONDARY OUTCOMES:
Percentage of subjects who obtain funding for the submitted proposal | 30 Months
Institute-specific percentile of the priority score | 30 Months
Percentage of subjects who submit proposals for funding | 30 Months
Percentage of subjects who received a good score (<40 or <200) which may be associated with future funding of a resubmission | 30 Months
Percentage of subjects who obtained any career development award funding | 30 Months

CONTACTS AND LOCATIONS:
Overall Officials: Alka Kanaya, MD, Principal Investigator — University of California, San Francisco; Peter Bacchetti, PhD, Study Director — University of California, San Francisco; Clay Johnston, MD, PhD, Study Director — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States